CLINICAL TRIAL: NCT01076543
Title: Phase I/II Investigation of Temsirolimus Plus Lenalidomide in Relapsed Non-Hodgkin Lymphomas
Brief Title: Lenalidomide and Temsirolimus in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01456; NCI-2011-01456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-443-A; CDR0000666432; 8309 (Other: University of Chicago Comprehensive Cancer Center); 8309 (Other: CTEP); N01CM00071 (NIH); N01CM62201 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: AIDS-Related Hodgkin Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Follicular Lymphoma; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Waldenstrom Macroglobulinemia | interventions — Lenalidomide; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (lenalidomide, temsirolimus) (Experimental): Patients receive lenalidomide PO on days 1-21 and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 2 courses may continue therapy for up to 52 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Drug: Temsirolimus

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase I/II trial studies the side effects and the best dose of lenalidomide when given together with temsirolimus and to see how well it works in treating patients with Hodgkin lymphoma or non-Hodgkin lymphoma that has come back after a period of improvement or is not responding to treatment. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Lenalidomide may also stop the growth of Hodgkin lymphoma or non-Hodgkin lymphoma by blocking blood flow to the cancer. Temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving lenalidomide together with temsirolimus may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, toxicity, and maximum tolerated dose of lenalidomide when combined with temsirolimus in patients with relapsed lymphomas. (Phase I) II. To determine complete and overall response rate of lenalidomide plus temsirolimus in patients with relapsed lymphomas as stratified by histology: follicular lymphoma, diffuse large B-cell lymphoma, and lymphoma not otherwise specified (NOS) (including Hodgkin lymphoma, T-cell non-Hodgkin lymphoma [T-NHL], lymphoplasmacytic lymphoma, and mantle cell lymphoma). (Phase II) III. To determine duration of response, progression-free survival, and overall survival of lenalidomide plus temsirolimus in patients with relapsed lymphomas as stratified by histology: diffuse large B-cell lymphoma, follicular lymphoma, and lymphoma NOS (including Hodgkin lymphoma, T-NHL, lymphoplasmacytic lymphoma, mantle cell lymphoma). (Phase II)

SECONDARY OBJECTIVES:

I. To determine mammalian target of rapamycin (mTOR) pathway activation in pre-treatment tumor tissue.

II. To determine angiogenic and microenvironmental status of pre-treatment tissue and peripheral blood samples, and to evaluate changes following treatment with temsirolimus and lenalidomide.

III. To determine differentially expressed genes associated with differences in clinical response and in progression-free survival (PFS) in patients with diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL) (Groups A and B, respectively).

IV. To determine a methylation signature predictive of clinical response and PFS in patients with DLBCL and FL (Groups A and B, respectively).

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Patients receive lenalidomide orally (PO) on days 1-21 and temsirolimus intravenously (IV) over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 2 courses may continue therapy for up to 52 weeks.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histology: bone marrow biopsies (with the exception of lymphoplasmacytic lymphoma) as the sole means of diagnosis are not acceptable; fine needle aspirates are not acceptable

  * Phase I: previously treated, histologically confirmed Hodgkin and non-Hodgkin lymphomas; the only exception to a requirement for a lymph node biopsy is lymphoplasmacytic lymphoma, which can be diagnosed based on morphologic evidence in the bone marrow plus the appropriate paraprotein
  * Phase II: previously treated, histologically confirmed mature non-Hodgkin lymphoma (NHL) stratified by histology:

    * Group A: diffuse large B-cell lymphoma (NOTE: all patients with DLBCL must have germinal center vs. non-germinal center phenotype established via immunohistochemistry)
    * Group B: follicular lymphoma
    * Group C: lymphoma NOS (including Hodgkin lymphoma, T-NHL, marginal zone lymphoma, lymphoplasmacytic
* No limit to number of prior therapies; prior autologous transplantation is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelet count >= 75,000/uL
* Total bilirubin =< 1.5 times upper limit of normal (ULN) (unless due to Gilbert's)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times ULN
* Creatinine clearance >= 60 mL/min as determined by calculated Cockcroft-Gault equation
* Fasting serum cholesterol =< 350 mg/dL
* Fasting serum triglycerides =< 2.5 times ULN
* All patients are required to have measurable disease; non-measurable disease alone is not acceptable; any tumor mass > 1 cm is acceptable; lesions that are considered non-measurable include the following:

  * Bone lesions (lesions if present should be noted)
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Bone marrow (involvement by lymphoma should be noted)
  * For Waldenstrom's macroglobulinemia, measurable disease is defined as at least one lesion with a single diameter of greater than 2 cm by computed tomography or bone marrow involvement with greater than 10% malignant cells and quantitative monoclonal protein (immunoglobulin M [IgM], IgG, IgA) greater than 1,000 mg/dL
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Ability to understand and the willingness to sign a written informed consent document
* Patients who are human immunodeficiency virus (HIV) positive are allowed to participate BUT must meet the following criteria:

  * No acquired immune deficiency syndrome (AIDS)-defining illness, AND
  * Cluster of differentiation (CD) 4 count >= 400 cells/mm^3, AND
  * No anti-retroviral therapy (including high-active antiretroviral therapy [HAART]) within 7 days of starting protocol therapy, AND
  * Patient may not take concurrent anti-retroviral therapy (including HAART) while on protocol
  * NOTE: it is not generally recommended to suspend anti-retroviral therapy (including HAART); the medical team enrolling a patient who suspends anti-retroviral therapy for the purpose of study participation must have a documented note reviewing the potential risks/benefits with the patient in the medical chart

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biological composition to temsirolimus or lenalidomide used in study
* Patients requiring active anti-retroviral therapy for HIV are excluded
* No "currently active" second malignancy, other than non-melanoma skin cancers; patients are not considered to have a "currently active" second malignancy if they have completed anti-cancer therapy and are considered by their physicians to be at less than 30% risk of relapse
* No history (within 3 months of study entry) of deep venous thrombosis/pulmonary embolism (DVT/PE); patients with a distant history (greater than 3 months before study entry) of DVT/PE are eligible, but should receive prophylactic aspirin or low molecular weight heparin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with relapsed/refractory DLBCL or HL who are eligible and willing to undergo potentially curative stem cell transplant
* Patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) are excluded
* No corticosteroids within 14 days prior to study, except for maintenance therapy for a non-malignant disease; maintenance therapy dose may not exceed 10 mg/day prednisone or equivalent; any patient on steroid therapy must receive thromboembolic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-04-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (11):
- United States (11):
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mercy Hospital Saint Louis, St Louis, Missouri

REFERENCES:
- [Derived] Major A, Kline J, Karrison TG, Fishkin PAS, Kimball AS, Petrich AM, Nattam S, Rao K, Sleckman BG, Cohen K, Besien KV, Rapoport AP, Smith SM. Phase I/II clinical trial of temsirolimus and lenalidomide in patients with relapsed and refractory lymphomas. Haematologica. 2022 Jul 1;107(7):1608-1618. doi: 10.3324/haematol.2021.278853. PMID 34320785

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, All Histologies, Lenalidomide 15 mg: Patients receive lenalidomide 15 mg PO on days 1-21 and 25 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. .
- Phase I, All Histologies, Lenalidomide 20 mg; Phase II, Diffuse Large B-Cell Subtype; Phase II, Lymphoma NOS: Patients receive lenalidomide 20 mg PO on days 1-21 and 25 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. .
- Phase I, All Histologies, Lenalidomide 25 mg: Patients receive lenalidomide 25 mg PO on days 1-21 and 25 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. .
- Phase II, Follicular Subtype: Patients receive lenalidomide 20mg PO on days 1-21 and 25 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. .
Period: Overall Study
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS
Started | 8 | 3 | 6 | 39 | 15 | 39
Completed | 6 | 3 | 6 | 39 | 15 | 39
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I, All Histologies, Lenalidomide 15 mg: Patients receive lenalidomide 15 mg PO on days 1-21 and25 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. .
- Total: Total of all reporting groups
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS | Total
Number analyzed (Participants) | 8 | 3 | 6 | 39 | 15 | 39 | 110
Age, Continuous [Mean (Full Range); unit: years] | 60.9 [41 to 73] | 65.2 [56 to 77] | 65.3 [41 to 80] | 64.1 [25 to 78] | 63.3 [43 to 76] | 47.4 [23 to 72] | 57.9 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 11 | 6 | 14 | 36
  Male | 7 | 2 | 3 | 28 | 9 | 25 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 4 | 2 | 6 | 14
  White | 8 | 1 | 5 | 33 | 12 | 29 | 88
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 6 | 39 | 15 | 39 | 110

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicity (DLT), Phase I Patients Only
Description: Incidence of dose-limiting toxicity (DLT) defined as any grade 3 or 4 adverse events as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I)
Time Frame: 28 days
Population: Only phase I patients were assessed for dose-limiting toxicity per 3+3 dose-escalation design to determine the maximum tolerated dose (MTD).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS
Number analyzed (Participants) | 6 | 3 | 6 | 0 | 0 | 0
Participants | 1 | 0 | 3 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Phase I, All Histologies, Lenalidomide 15 mg vs Phase I, All Histologies, Lenalidomide 20 mg vs Phase I, All Histologies, Lenalidomide 25 mg; Test type: Other; Maximum tolerated dose in mg = 20 — The maximum tolerated dose (MTD) was determined using the traditional "3+3" design and was the maximum dose level such that less than 33% of the patients (i.e, <1 of 3 or <2 of 6) experience dose-limiting toxicity

2. Primary Outcome: Complete Response (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions;
Time Frame: Up to 1 year
Population: Only phase II patients were assessed for complete response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS
Number analyzed (Participants) | 0 | 0 | 0 | 39 | 15 | 39
Participants | 0 | 0 | 0 | 5 | 5 | 7

3. Primary Outcome: Overall Response Rate (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Population: Only phase II patients were assessed for overall response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS
Number analyzed (Participants) | 0 | 0 | 0 | 39 | 15 | 39
Participants | 0 | 0 | 0 | 10 | 7 | 25
Statistical Analysis 1: Comparison: Phase II, Diffuse Large B-Cell Subtype; Two-stage, minimax design was used to test the null hypothesis that the overall response rate was 30% vs. a 50% alternative; Test type: Superiority; p > 0.10, Binomial exact test; The number of responders required to reject the null hypothesis was 16 or more
Statistical Analysis 2: Comparison: Phase II, Follicular Subtype; Two-stage, minimax design was used to test the null hypothesis that the overall response rate was 50% vs. 70% alternative; Test type: Superiority; The follicular subgroup did not reach its accrual goal and was closed
Statistical Analysis 3: Comparison: Phase II, Lymphoma NOS; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.10, Binomial exact test; The number of responders required to reject the null hypothesis was 16 or more

4. Secondary Outcome: Progression-free Survival (PFS) (Phase II)
Description: Kaplan-Meier curves will be generated for PFS stratified by histology; median PFS times will be determined and 90% confidence intervals derived as described in Brookmeyer and Crowley.
Time Frame: Time from study entry until disease progression or death from any cause, assessed up to 5 years
Population: Note: Only phase II patients were followed for progression-free survival.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS
Number analyzed (Participants) | 0 | 0 | 0 | 39 | 15 | 39
Months |  |  |  | 7.0 [3.5 to 8.0] | 27.7 [6.5 to 35.8] | 7.0 [4.6 to 9.9]

5. Secondary Outcome: Overall Survival (OS) (Phase II)
Description: Kaplan-Meier curves will be generated for OS stratified by histology; median OS times will be determined and 90% confidence intervals derived as described in Brookmeyer and Crowley.
Time Frame: Time from study entry until death from any cause, assessed up to 6 years
Population: Only phase II patients were followed for overall survival.
  Note:999999 for the upper confidence interval of the median for the follicular subtype means "not estimable."
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS
Number analyzed (Participants) | 0 | 0 | 0 | 39 | 15 | 39
Months |  |  |  | 9.1 [6.0 to 16.0] | 35.8 [18.8 to NA] — The upper confidence limit could not be determined due to the censoring. | 25.5 [10.8 to 60.6]

ADVERSE EVENTS:
Time Frame: Mortality collected up to 6 years; all other AEs collected up to 2 years.
Arm/Group | Phase I, All Histologies, Lenalidomide 15 mg | Phase I, All Histologies, Lenalidomide 20 mg | Phase I, All Histologies, Lenalidomide 25 mg | Phase II, Diffuse Large B-Cell Subtype | Phase II, Follicular Subtype | Phase II, Lymphoma NOS
All-Cause Mortality (participants affected / at risk) | 4/8 | 3/3 | 4/6 | 23/39 | 4/15 | 18/39
Serious Adverse Events (participants affected / at risk) | 2/8 | 2/3 | 5/6 | 22/39 | 7/15 | 22/39
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 6/6 | 39/39 | 13/15 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, All Histologies, Lenalidomide 15 mg (N=8) | Phase I, All Histologies, Lenalidomide 20 mg (N=3) | Phase I, All Histologies, Lenalidomide 25 mg (N=6) | Phase II, Diffuse Large B-Cell Subtype (N=39) | Phase II, Follicular Subtype (N=15) | Phase II, Lymphoma NOS (N=39)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 8 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Vascular disorders - other (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 2 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
INR increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mood alteration - depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous disorders - other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis/Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colonic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Surgical and medical procedures - other (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, All Histologies, Lenalidomide 15 mg (N=8) | Phase I, All Histologies, Lenalidomide 20 mg (N=3) | Phase I, All Histologies, Lenalidomide 25 mg (N=6) | Phase II, Diffuse Large B-Cell Subtype (N=39) | Phase II, Follicular Subtype (N=15) | Phase II, Lymphoma NOS (N=39)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 9 | 1 | 7
Alkaline aminotransferase increase (Investigations) | 4 | 1 | 2 | 12 | 7 | 21
Alkaline phosphatase increased (Investigations) | 2 | 1 | 1 | 9 | 6 | 17
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3 | 2 | 5
Anemia (Blood and lymphatic system disorders) | 7 | 2 | 4 | 33 | 10 | 36
Anorexia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 20 | 8 | 18
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 1 | 15 | 6 | 20
Bleeding (Blood and lymphatic system disorders) | 2 | 0 | 0 | 7 | 2 | 9
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 2
Chills (General disorders) | 2 | 0 | 1 | 5 | 2 | 9
Cholesterol high (Investigations) | 4 | 1 | 1 | 11 | 3 | 16
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 17 | 8 | 18
Creatinine increased (Investigations) | 1 | 0 | 0 | 10 | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 12 | 6 | 14
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 2 | 14 | 4 | 14
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 6 | 4 | 6
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2 | 4 | 2 | 6
Dysgeusia (Nervous system disorders) | 2 | 1 | 2 | 9 | 7 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 6 | 6 | 6
Edema limbs (General disorders) | 2 | 2 | 1 | 9 | 8 | 8
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 1 | 4 | 25 | 12 | 31
Fever (General disorders) | 1 | 0 | 0 | 11 | 3 | 17
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2 | 1
Flushing (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 2 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3 | 3 | 29 | 9 | 33
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 2 | 0 | 2
Hypernatremia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 8 | 1 | 5
Hypertension (Vascular disorders) | 1 | 0 | 0 | 10 | 3 | 8
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 15 | 4 | 20
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 3 | 4 | 12 | 4 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3 | 3 | 23 | 6 | 24
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3 | 2 | 23 | 7 | 30
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 12 | 1 | 11
Infection (Infections and infestations) | 1 | 0 | 0 | 6 | 2 | 3
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 6 | 3 | 7
Localized edema (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 1 | 9
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 5 | 2 | 2 | 28 | 10 | 31
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 12 | 4 | 12
Neck edema (General disorders) | 1 | 0 | 0 | 1 | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 2 | 2 | 1 | 6 | 5 | 8
Neutrophil count decreased (Investigations) | 5 | 2 | 3 | 28 | 9 | 26
Pain (General disorders) | 2 | 0 | 2 | 14 | 6 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 4 | 2 | 3
Platelet count decreased (Investigations) | 7 | 2 | 5 | 32 | 12 | 32
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 12 | 6 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 18 | 8 | 14
Rash/dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 12 | 4 | 8
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 1
Sinus pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 3 | 4 | 2
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 3
Skin infection (Infections and infestations) | 1 | 0 | 0 | 5 | 1 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 7 | 2 | 6
White blood cell decreased (Investigations) | 5 | 3 | 5 | 32 | 10 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4 | 2 | 2
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 6 | 1 | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 9 | 2 | 11
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 2 | 4 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 3 | 1
Gum infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hypothryoidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 7 | 2 | 3
Nervous system disorders - other (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 7
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 8 | 1 | 8
Stomatitis/pharyngitis (Infections and infestations) | 0 | 0 | 1 | 7 | 4 | 11
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 4 | 3 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 3 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 4 | 2 | 7
Cataract (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 2
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 1
Edema face (General disorders) | 0 | 0 | 0 | 3 | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 7 | 2 | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 1 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 5 | 2 | 7
INR increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 3
Mood alteration - depression (Psychiatric disorders) | 0 | 0 | 0 | 3 | 1 | 3
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 5
Non-cardiac chest pain (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 3 | 3
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 4
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 3
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 2 | 3 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3 | 5
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Neuropathy - motor (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Edema trunk (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 2
Injury, poisoning and procedural complications - other (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Investigations - other (Investigations) | 0 | 0 | 0 | 1 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Tooth development disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT01076543/Prot_SAP_000.pdf